CLINICAL TRIAL: NCT05699291
Title: Analysis of the Cost of Using FLUOrescence in Green of Indocyanine for the Detection of the Sentinel Lymph Node in the Breast Cancer.
Brief Title: Cost of Using FLUOrescence to Green of Indocyanine for the Detection of Breast Cancer.
Acronym: FLUOBREAST-2
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02271-42
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Sentinel Lymph Node

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient eligible for the sentinel lymph node technique by lndocyanine Green.: To evaluate the overall cost at 1 month of the sentinel lymph node detection technique using Indocyanine Green in patients with breast cancer, from the point of view of the health insurance and the hospital.
  Interventions: Other: Sentinel node detection technique
- Patient eligible for the sentinel lymph node technique by isotopes.: To evaluate the overall cost at 1 month of the sentinel lymph node detection technique using isotopes in patients with breast cancer, from the point of view of health insurance and the hospital.
  Interventions: Other: Sentinel node detection technique

INTERVENTIONS:
Other: Sentinel node detection technique — Patients cared for by a surgeon for histologically proven breast cancer and for whom an indication for detection of the sentinel lymph node is posed.

SUMMARY:
The purpose of this study is to analyze the average direct costs of each of these techniques, represented by the costs directly linked to the management of breast cancer, to the surgical intervention and to the techniques evaluated (Indocyanine Green and isotopes) which are: consultations, hospitalizations, resources consumed during the surgical intervention, as well as the time of the patients, transport...

DETAILED DESCRIPTION:
The main objective is to evaluate the overall cost at 1 month of the sentinel lymph node detection technique using Indocyanine Green compared to the technique using isotopes in patients with breast cancer, from the point of view of health insurance and the hospital.

The chosen time horizon is up to 1 month post-intervention. The choice of this time horizon corresponds to the usual duration of follow-up for patients who have benefited from one of the sentinel lymph node detection techniques, in order to collect the main post-surgical complications.

This is a multicenter, prospective, observational, non-randomized study, aimed at comparing the overall cost of two sentinel lymph node detection techniques (Indocyanine Green and isotope) from a dual perspective (health insurance and hospital).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over, having given her oral non-objection ;
* Patient with histologically proven breast cancer ;
* Patient eligible for the sentinel lymph node technique by Indocyanine Green or isotopes.

Exclusion Criteria:

* Patient who has expressed her opposition to the use of her medical data ;
* Patient under legal protection, guardianship or curatorship ;
* Pregnant patient ;
* Patient not affiliated to a social security scheme.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with histologically proven breast cancer
Study Population: Patient with histologically proven breast cancer, eligible for sentinel lymph node technique by Indocyanine Green or isotopes
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Average direct costs of the two techniques assessed (Indocyanine Green and isotopes) | 1 month
  To evaluate the overall cost at 1 month of the sentinel lymph node detection technique using Indocyanine Green compared to the technique using isotopes in patients with breast cancer, from the point of view of the health insurance and the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé des Peupliers, Paris, France

IPD SHARING:
Plan to Share IPD: No